CLINICAL TRIAL: NCT00241748
Title: Pharmacoepidemiology and Pharmacogenetics of a Statin Adverse Event
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bruce Psaty, Professor, University of Washington
Other Study IDs: 1310; R01HL078888 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Rhabdomyolysis
MeSH Terms: conditions — Rhabdomyolysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA is extracted from swish and spit samples. DNA is retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Rhabdomyolysis Case Subjects
- 2: Heart and Vascular Health Study statin users - control group 1
- 3: Cardiovascular Health Study statin users - control group 2

SUMMARY:
To conduct a case-control study of factors that increased the risk of rhabdomyolysis, an adverse drug reaction in cerivastatin users

DETAILED DESCRIPTION:
BACKGROUND:

Cerivastatin (Baycol), an HMG-CoA reductase inhibitor (statin), was approved and marketed in early 1998 for the treatment of dyslipidemias. Soon afterwards, suspected adverse drug reaction (SADR) reports in cerivastatin users often cited rhabdomyolysis, an uncommon condition in which the breakdown of skeletal muscle cells causes pain, weakness and, in-some cases, renal failure or death. By the time that cerivastatin was withdrawn from the market in 2001, the FDA had received 1,899 SADRs for rhabdomyolysis associated with cerivastatin compared to 1,440 for all other statins combined. In an analysis conducted by FDA scientists, the relative reporting rate (RRR) of fatal rhabdomyolysis was 40 times higher among users of cerivastatin than among users of other statins. For the outcome of all fatal and non-fatal rhabdomyolysis, the RRR was 54 times higher. About half of the rhabdomyolysis cases occurred in subjects who had taken both cerivastatin and gemfibrozil. Subsequently, pharmacokinetic studies demonstrated that gemfibrozil inhibits both major metabolic pathways for cerivastatin-not only the Cytochrome P-450 (CYP) 2C8-mediated oxidation, but also the glucuronidation by uridine diphosphate glucuronysyltransferases (UGT). The investigators hypothesize that rhabdomyolysis cases who were taking cerivastatin but not gemfibrozil had one or both of two types of risk factors: (1) medications that are known inhibitors of these enzymes; or (2) functional genetic variants in one or more of the CYP or UGT enzymes.

Coronary heart disease (CHD) is the leading cause of morbidity and mortality in the U.S. and statin agents are commonly employed for the treatment of hyperlipidemia, one of the principal risk factors for CHD. Given the hundreds of thousands to millions of Americans presently on statin therapy, and the potentially serious (though relatively rare) complication of rhabdomyolysis, this is a significant topic to study.

DESIGN NARRATIVE:

The investigators hypothesize that rhabdomyolysis cases who were taking cerivastatin but not gemfibrozil had one or both of two types of risk factors: (1) medications that are known inhibitors of these enzymes; or (2) functional genetic variants in one or more of the CYP or UGT enzymes. This project is a case-control study of factors that increased the risk of rhabdomyolysis in cerivastatin users. Cases will be cerivastatin users who had rhabdomyolysis, and statin users from two on-going epidemiologic studies will serve as two complementary control groups. "For cases, identified with the assistance of attorneys, a review of medical records and telephone interview will verify the diagnosis and provide information on medication use. Subjects will also return a mouthwash buccal sample for DNA extraction. All subjects will be genotyped for known functional variants in CYP2C8, UGT1A1 and UGT1A3. In the hypothesis-testing part of this case-control study, medications known to be inhibitors of these enzymes and functional variants in their genes will be evaluated as risk factors for rhabdomyolysis in cerivastatin users. Additionally, pharmacoepidemiologic analyses of the FDA AERS data will be conducted to identify other potential new drug-drug interactions. Power to detect expected effect sizes is 80% or greater. In the discovery phase of the project, the DNA of rhabdomyolysis cases who did not take gemfibrozil will be sequenced to identify new single nucleotide polymorphisms (SNPs) in CYP2C8, UGT1 Al and UGT1 A3. The functional significance of new pharmacoepidemiologic associations will be evaluated in in vitro pharmacokinetic inhibition studies. Additionally, newly discovered SNPs in CYP2C8 will be expressed in E. coli and evaluated for their functional significance.

ELIGIBILITY:
Inclusion Criteria:

* Older than 30 years old

Exclusion Criteria:

* Recent history of trauma

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases: persons suffering cervistatin-associated rhabdomyolysis who sued the manufactorer and settled their case Control 1: statin users participating in the Heart and Vascular Health Study Control 2: statin users participating in the Cardiovascular Health Study
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2005-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce M Psaty, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States